CLINICAL TRIAL: NCT04921241
Title: In Utero Exposure to SARS-CoV-2 (COVID-19) and Cardiovascular and Metabolic Endpoints in Early Life
Acronym: PROSPER
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lindsay Fourman, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2021P001107
Record Dates: First submitted 2021-06-07; First posted 2021-06-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: In Utero SARS-CoV-2 Exposure
Keywords: metabolic disease; cardiovascular disease
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 Exposed Dyads: Mothers who had SARS-CoV-2 during pregnancy and their offspring
  Interventions: Other: In Utero Exposure to SARS-CoV-2
- SARS-CoV-2 Unexposed Dyads: Mothers who were not known to have SARS-CoV-2 during pregnancy and their offspring

INTERVENTIONS:
Other: In Utero Exposure to SARS-CoV-2 — Born to mother with SARS-CoV-2 infection during pregnancy
  Groups: SARS-CoV-2 Exposed Dyads

SUMMARY:
Since its initial outbreak in late 2019, coronavirus disease 2019 (COVID-19) caused by the novel coronavirus SARS-CoV-2 has ravaged the globe, causing illness characterized by inflammation and impaired oxygen levels. As a particularly vulnerable group, pregnant women have had a heightened prevalence and severity of infection. In this context, a new population of children has emerged who were exposed to maternal COVID-19 in the womb. As maternal diseases during pregnancy may impact the health of offspring over the life course, health outcomes among these individuals must be urgently evaluated. In the current study, the investigators will leverage a perinatal biorepository comprised of pregnant women with and without COVID-19 to delineate the metabolic and cardiovascular risk profiles of these offspring. This work stands to benefit the burgeoning population of children exposed to COVID-19 in the womb and to deepen the mechanistic understanding of developmental origins of cardiometabolic disease with respect to maternal infections.

ELIGIBILITY:
Inclusion Criteria:

* Mother with or without prenatal COVID-19 who was enrolled in the MGH COVID-19 Perinatal Biorepository and her child (9-24 months old)

Exclusion Criteria:

* Child with any history of documented COVID-19
* Mother who received the COVID-19 vaccine during pregnancy with her child
* Significant chronic illness in mother or child judged by the investigator to represent a contraindication to study participation

Min Age: 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We are recruiting mothers who had COVID-19 during pregnancy and their offspring (9-24 months old). We are also recruiting mothers who were at risk for but not infected with COVID-19 during pregnancy and their children to serve as controls. Mothers in both arms had been contemporaneously enrolled in the MGH COVID-19 Perinatal Biorepository during pregnancy.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Aortic pulse-wave velocity | Baseline

SECONDARY OUTCOMES:
Skinfold thicknesses (subscapular, triceps) | Baseline
Weight-for-length z-score | Baseline
Systolic and diastolic blood pressure | Baseline
Beta index of aortic stiffness using echocardiogram | Baseline
Aortic intima-media thickness using echocardiogram | Baseline
Urinary angiotensin peptide levels | Baseline
Urinary angiotensin converting enzyme (ACE) levels | Baseline
Left ventricular mass | Baseline
Left ventricular dimensions | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States